CLINICAL TRIAL: NCT06454838
Title: Exercise Capacity Muscle Oxygenation and Arterial Stiffness in Children With Pulmonary Arterial Hypertension
Status: Recruiting | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Meral Boşnak Güçlü, Prof. Dr., Gazi University
Other Study IDs: Gazi University 2024
Record Dates: First submitted 2024-05-20; First posted 2024-06-12 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Upper Extremity Exercise Capacity; Muscle Oxygenation; Arterial Stiffness; Respiratory Muscle Strength
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with pulmonary arterial hypertension: Pulmonary function (spirometer), respiratory muscle strength (mouth pressure device), upper extremity exercise capacity (Six minutes PegBoard Ring Test) and lower extremity exercise capacity (Six minutes walk test), muscle oxygenation ('Moxy' monitor device), dyspnea (modified Borg Scale), peripheral muscle strength (hand-held dynamometer), arterial stiffness (arteriograph), physical activity level (multi-sensor activity monitor) and static balance (balance system with computed) will be evaluated.
- Age- and sex- matched healthy controls: Pulmonary function (spirometer), respiratory muscle strength (mouth pressure device), upper extremity exercise capacity (Six minutes PegBoard Ring Test) and lower extremity exercise capacity (Six minutes walk test), muscle oxygenation ('Moxy' monitor device), dyspnea (modified Borg Scale), peripheral muscle strength (hand-held dynamometer), arterial stiffness (arteriograph), physical activity level (multi-sensor activity monitor) and static balance (balance system with computed) will be evaluated.

SUMMARY:
The primary aim is to evaluate pulmonary function, respiratory muscle strength, upper and lower extremity exercise capacity, muscle oxygenation, dyspnea, peripheral muscle strength, arterial stiffness, physical activity level and balance in children with pulmonary arterial hypertension and compare with age- and sex-matched healthy controls.

The second aim is to investigate the relationship between upper extremity exercise capacity, arterial stiffness, respiratory and peripheral muscle strength

DETAILED DESCRIPTION:
Pulmonary arterial hypertension (PAH) is defined as higher than 25 mmHg in mean pulmonary arterial pressure at rest. Pulmonary arterial hypertension is chronic and progressive disease.

Symptoms such as dyspnea, fatigue, exercise intolerance, cyanosis and syncope are shown in children with PAH. Most common symptom is dyspnea during exertion. Dyspnea at rest could occur while the severity of disease is progressed. All these symptoms have been associated with decreased cardiac output and mismatch oxygen transport.

This study is planned as a cross-sectional study. At least 13 children with PAH and at least 13 age- and sex- matched healthy controls will be included in this study. Individuals' pulmonary function (spirometer), respiratory muscle strength (mouth pressure device), upper extremity exercise capacity (the six minute Peg Board Ring Test), lower extremity exercise capacity (six minute walk test), muscle oxygenation ('Moxy' monitor device), dyspnea (modified Borg Scale), peripheral muscle strength (hand-held dynamometer), arterial stiffness (arteriograph device), physical activity level (multi-sensor activity monitor) and static balance (balance system with computed) will evaluated in children with PAH and healthy controls. All assessments will be completed in two days.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Between the ages of 6-18
* Diagnosed with pulmonary arterial hypertension
* Stability of clinical condition and receiving standard medical treatment

Healthy controls:

* Between the ages of 6-18
* Willing to participate in the study

Exclusion Criteria:

Patients:

* Having any acute infection, orthopedic, neurological, cooperation, vision or hearing problems that may prevent during the measurements
* Participated in a planned exercise program in a last three months

Healthy controls:

* Having any acute or chronic illness
* Active or ex-smoker

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: At least 13 children with PAH and 13 age- and sex- matched healthy controls will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Estimated)
Dates: Start 2024-04-30 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Upper extremity exercise capacity | First day
  Six minutes PegBoard and Ring Test (6-PBRT) will be applied to evaluate upper extremity exercise capacity. There are a total of 20 rings and 2 wooden bars at above and 2 wooden bars at below. Patients will be asked to move the each two rings from upper bars to lower bars and than from lower bars to upper bars with hands as fast as.
  The total number of rings moved during the test will be recorded at the end of test.
Muscle oxygenation | First day
  Muscle oxygenation will be evaluated with the Moxy monitor (Moxy, Fortiori Design LLC, Minnesota, USA) as a non-invasive. The device will be attached with soft tape on the participants' skin surface.
  The device will be placed on the 1/3 lower motor point of the deltoid muscle group of the dominant arm during the the six minutes PegBoard and Ring Test and placed on the 1/3 lower motor point of the quadriceps muscle of dominant leg during the six minutes walk test. At rest and during the test, skeletal muscle oxygenation (StO2) and total hemoglobin (THb) values will be recorded.

SECONDARY OUTCOMES:
Respiratory muscle strength | First day
  Maximal inspiratory (MIP) and maximal expiratory (MEP) pressures expressing respiratory muscle strength will be evaluated using a portable mouth pressure device. Measurements will be applied according to American Thoracic Society and European Respiratory Society criteria.
Peripheral muscle strength | Second day
  Isometric peripheral muscle strength of quadriceps and deltoid muscles will be measured with a portable hand-held dynamometer (JTECH Commander, USA). Measurements will be repeated three times for both extremities.
Dyspnea | Second day
  Perception of dyspnea at rest and during the activities of daily living will be assessed with modified Borg scale. The scale is graded between '0' and '10'. The lower score for dyspnea means 'no shortness of breath' and higher score for dyspnea means 'very very hard'.
Lower extremity exercise capacity | Second day
  Six minute walk test (6-MWT) will be used to evaluate lower extremity exercise capacity. The test will be applied based on American Thoracic Society and European Respiratory Society criteria. The longest walking distance will be recorded to analyze.
Physical activity (Total energy expenditure) | Second day
  Total energy expenditure, one of the parameters of physical activity, will be evaluated with multisensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient will wear the multisensor physical activity monitor over the triceps muscle of the right arm for 3 continuous days. Total energy expenditure will be expressed as joule/day. The parameter measured over two days will be averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical activity (Active energy expenditure) | Second day
  Active energy expenditure, one of the parameters of physical activity, will be evaluated with multisensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient will wear the multisensor physical activity monitor over the triceps muscle of the right arm for 3 continuous days. Active energy expenditure will be expressed as joule/day. The parameter measured over two days will be averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical activity (Physical activity duration) | Second day
  Physical activity duration, one of the parameters of physical activity, will be evaluated with multisensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient will wear the multisensor physical activity monitor over the triceps muscle of the right arm for 3 continuous days. Physical activity duration will be expressed as minute/day. The parameter measured over two days will be averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical activity (Average metabolic equivalent) | Second day
  Average metabolic equivalent, one of the parameters of physical activity, will be evaluated with multisensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient will wear the multisensor physical activity monitor over the triceps muscle of the right arm for 3 continuous days. The parameter measured over two days will be averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical activity (Number of steps) | Second day
  Number of steps, one of the parameters of physical activity, will be evaluated with multisensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient will wear the multisensor physical activity monitor over the triceps muscle of the right arm for 3 continuous days. Number of steps will be expressed as steps/day. The parameter measured over two days will be averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical activity (Lying down duration) | Second day
  Lying down duration, one of the parameters of physical activity, will be evaluated with multisensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient will wear the multisensor physical activity monitor over the triceps muscle of the right arm for 3 continuous days. Lying down duration will be expressed as minutes/day. The parameter measured over two days will be averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical activity (Sleep duration) | Second day
  Sleep duration, one of the parameters of physical activity, will be evaluated with multisensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient will wear the multisensor physical activity monitor over the triceps muscle of the right arm for 3 continuous days. Sleep duration will be expressed as minutes/day. The parameter measured over two days will be averaged and analyzed with the "SenseWear® 7.0 Software" program.
Pulmonary function (Forced expiratory volume in the first second (FEV1)) | First day
  Pulmonary function will be evaluated with the spirometry based on American Thoracic Society and European Respiratory Society criteria. Forced expiratory volume in the first second (FEV1) will be measured.
Pulmonary function (Forced vital capacity (FVC)) | First day
  Pulmonary function will be evaluated with the spirometry based on American Thoracic Society and European Respiratory Society criteria. Forced vital capacity (FVC) will be measured.
Pulmonary function (FEV1 / FVC) | First day
  Pulmonary function will be evaluated with the spirometry based on American Thoracic Society and European Respiratory Society criteria. FEV1/FVC will be measured.
Pulmonary function (Peak flow rate (PEF)) | First day
  Pulmonary function will be evaluated with the spirometry based on American Thoracic Society and European Respiratory Society criteria. Peak flow rate (PEF) will be measured.
Pulmonary function (Flow rate 25-75% of forced expiratory volume (FEF 25-75%)) | First day
  Pulmonary function will be evaluated with the spirometry based on American Thoracic Society and European Respiratory Society criteria. Flow rate 25-75% of forced expiratory volume (FEF 25-75%) will be measured.
Balance | Second day
  Static balance will be evaluated using a balance assessment device.
Arterial Stiffness | Second day
  Arterial stiffness will be assessed non-invasively with arteriography device. Carotid-femoral artery pulse wave velocity, augmented index, systolic and diastolic pressures and mean arterial pressures of aort and brachial arteries will be measured. Carotid-femoral artery pulse wave velocity will be measured with tonometer on carotid artery and augmented index will be measured with sphygmomanometer on brachial artery.

CONTACTS AND LOCATIONS:
Overall Officials: Meral BOŞNAK GÜÇLÜ, Prof. Dr., Study Director — Gazi University; Ece BAYTOK, Pt. MSc., Study Chair — Gazi University; Betül YOLERİ, Pt. MSc., Principal Investigator — Gazi University; Fatma HAYVACI CANBEYLİ, M.D., Principal Investigator — Gazi University; Serdar KULA, Prof. Dr., Principal Investigator — Gazi University
Locations (1):
- Gazi University Faculty of Health Sciences Department of Physiotherapy and Rehabilitation, Cardiopulmonary Rehabilitation Unit, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holland AE, Spruit MA, Troosters T, Puhan MA, Pepin V, Saey D, McCormack MC, Carlin BW, Sciurba FC, Pitta F, Wanger J, MacIntyre N, Kaminsky DA, Culver BH, Revill SM, Hernandes NA, Andrianopoulos V, Camillo CA, Mitchell KE, Lee AL, Hill CJ, Singh SJ. An official European Respiratory Society/American Thoracic Society technical standard: field walking tests in chronic respiratory disease. Eur Respir J. 2014 Dec;44(6):1428-46. doi: 10.1183/09031936.00150314. Epub 2014 Oct 30. PMID 25359355
- [Background] Li AM, Yin J, Au JT, So HK, Tsang T, Wong E, Fok TF, Ng PC. Standard reference for the six-minute-walk test in healthy children aged 7 to 16 years. Am J Respir Crit Care Med. 2007 Jul 15;176(2):174-80. doi: 10.1164/rccm.200607-883OC. Epub 2007 Apr 26. PMID 17463419
- [Background] Feldmann A, Schmitz R, Erlacher D. Near-infrared spectroscopy-derived muscle oxygen saturation on a 0% to 100% scale: reliability and validity of the Moxy Monitor. J Biomed Opt. 2019 Nov;24(11):1-11. doi: 10.1117/1.JBO.24.11.115001. PMID 31741352
- [Background] Crum EM, O'Connor WJ, Van Loo L, Valckx M, Stannard SR. Validity and reliability of the Moxy oxygen monitor during incremental cycling exercise. Eur J Sport Sci. 2017 Sep;17(8):1037-1043. doi: 10.1080/17461391.2017.1330899. Epub 2017 May 30. PMID 28557670
- [Background] Beenakker EA, van der Hoeven JH, Fock JM, Maurits NM. Reference values of maximum isometric muscle force obtained in 270 children aged 4-16 years by hand-held dynamometry. Neuromuscul Disord. 2001 Jul;11(5):441-6. doi: 10.1016/s0960-8966(01)00193-6. PMID 11404114
- [Background] Rosenzweig EB, Abman SH, Adatia I, Beghetti M, Bonnet D, Haworth S, Ivy DD, Berger RMF. Paediatric pulmonary arterial hypertension: updates on definition, classification, diagnostics and management. Eur Respir J. 2019 Jan 24;53(1):1801916. doi: 10.1183/13993003.01916-2018. Print 2019 Jan. PMID 30545978
- [Background] Kula S, Canbeyli F, Atasayan V, Tunaoglu FS, Oguz AD. A retrospective study on children with pulmonary arterial hypertension: A single-center experience. Anatol J Cardiol. 2018 Jul;20(1):41-47. doi: 10.14744/AnatolJCardiol.2018.78370. PMID 29952362
- [Background] Zuk M, Migdal A, Jagiellowicz-Kowalska D, Mazurkiewicz K, Sadel-Wieczorek A, Brzezinska-Rajszys G. Six-Minute Walk Test in Evaluation of Children with Pulmonary Arterial Hypertension. Pediatr Cardiol. 2017 Apr;38(4):754-761. doi: 10.1007/s00246-017-1575-z. Epub 2017 Feb 27. PMID 28239753
- [Background] Atasayan V, Canbeyli F, Tunaoglu FS, Oguz AD, Celik B, Kula S. Prognostic value of oxygen saturation and heart rate during a six-minute walk test in pediatric pulmonary hypertension. Turk J Med Sci. 2021 Aug 30;51(4):1833-1840. doi: 10.3906/sag-2004-220. PMID 33754651